CLINICAL TRIAL: NCT01736241
Title: A Single-Dose, Dose-Escalation Study to Determine the Safety, Tolerability, and Pharmacokinetics of LY3053102 in Healthy Subjects
Brief Title: A Study of LY3053102 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 14514; I6I-MC-LMRA (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-11-26; First posted 2012-11-29 (Estimated); Results first posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2017-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY3053102 (Experimental): A single 2-, 7-, 20-, 50-, 150-, or 405-milligrams (mg) dose of LY3053102 was subcutaneously administered to newly randomized participants in 6 escalating dose level cohorts. The dose was escalated based on the safety results over at least a 7-day evaluation period postdose. The dose escalation occurred over 13 weeks proceeding according to tolerability at each dose level.
  Interventions: Drug: LY3053102
- Placebo (Placebo Comparator): A single dose of LY3053102-matching placebo was administered subcutaneously to 1 newly randomized participant in each LY3053102-dose level cohort over 13 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3053102
  Arms: LY3053102
Drug: Placebo
  Arms: Placebo

SUMMARY:
The main purpose of this study was to evaluate the safety and tolerability of the study drug known as LY3053102 in healthy participants. The study also investigated how much of the study drug entered the blood stream and how long it took the body to dispose of the study drug. Information about any side effects that occurred was also collected. The study was expected to last approximately 8 weeks for each participant (up to 4 weeks from screening to the administration of study drug and an additional 4 weeks of follow up).

ELIGIBILITY:
Inclusion Criteria:

* Normal blood pressure
* Female participants were not of child-bearing potential due to surgical sterilization (hysterectomy or bilateral oophorectomy or tubal ligation) or menopause
* Had a body mass index (BMI) of 18.5 to 40.0 kilograms per square meter (kg/m^2), inclusive, at screening

Exclusion Criteria:

* Had known allergies to LY3053102 or related compounds
* Had a history of significant disease that may have affected the actions of drugs or may pose a risk when taking the study medication
* Had a history of developing allergies, asthma, severe drug allergies (symptoms including, but not limited to, itching, red rashes, sores on the skin, scaling and shedding of skin), allergies or reactions to more than one drug, or have had bad reactions to skin creams containing corticosteroids
* Heavy smokers (more than 10 cigarettes a day)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-12; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Groups:
- 2 mg LY3053102: LY3053102: A single dose of 2 milligrams (mg), administered subcutaneously. The dose was escalated for a new cohort of randomized participants based on the safety results over at least a 7-day evaluation period postdose.
- 7 mg LY3053102: LY3053102: A single dose of 7 mg, administered subcutaneously. The dose was escalated for a new cohort of randomized participants based on the safety results over at least a 7-day evaluation period postdose.
- 20 mg LY3053102: LY3053102: A single dose of 20 mg, administered subcutaneously. The dose was escalated for a new cohort of randomized participants based on the safety results over at least a 7-day evaluation period postdose.
- 50 mg LY3053102: LY3053102: A single dose of 50 mg, administered subcutaneously. The dose was escalated for a new cohort of randomized participants based on the safety results over at least a 7-day evaluation period postdose.
- 150 mg LY3053102: LY3053102: A single dose of 150 mg, administered subcutaneously. The dose was escalated for a new cohort of randomized participants based on the safety results over at least a 7-day evaluation period postdose.
- 405 mg LY3053102: LY3053102: A single dose of 405 mg, administered subcutaneously.
- Placebo: Placebo: A single dose of LY3053102-matching placebo, administered subcutaneously to 1 newly randomized participant in each LY3053102-dose level cohort.
Period: Overall Study
Arm/Group | 2 mg LY3053102 | 7 mg LY3053102 | 20 mg LY3053102 | 50 mg LY3053102 | 150 mg LY3053102 | 405 mg LY3053102 | Placebo
Started | 6 | 6 | 6 | 5 | 6 | 6 | 6
Received at Least One Dose of Study Drug | 6 | 6 | 6 | 5 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 5 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | 2 mg LY3053102 | 7 mg LY3053102 | 20 mg LY3053102 | 50 mg LY3053102 | 150 mg LY3053102 | 405 mg LY3053102 | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.2 (9.7) | 33.2 (4.3) | 39.7 (11.1) | 36.2 (14.7) | 34.3 (10.7) | 31.0 (8.9) | 34.5 (7.4) | 34.8 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  Male | 5 | 6 | 5 | 5 | 6 | 6 | 6 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 41
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 6 | 5 | 5 | 5 | 6 | 5 | 38
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 3
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Singapore | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 41

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Adverse Events (AEs) or Any Serious AEs
Description: A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through Day 31
Population: Participants who received at least one dose of LY3053102 or placebo.
Measure: Number; unit: participants
Groups:
- 2 mg LY3053102: LY3053102: A single dose of 2 milligrams (mg), administered subcutaneously.
- 7 mg LY3053102: LY3053102: A single dose of 7 mg, administered subcutaneously.
- 20 mg LY3053102: LY3053102: A single dose of 20 mg, administered subcutaneously.
- 50 mg LY3053102: LY3053102: A single dose of 50 mg, administered subcutaneously.
- 150 mg LY3053102: LY3053102: A single dose of 150 mg, administered subcutaneously.
- Placebo: Placebo: A single dose of LY3053102-matching placebo, administered subcutaneously to 1 participant in each LY3053102-dose level cohort.
Arm/Group | 2 mg LY3053102 | 7 mg LY3053102 | 20 mg LY3053102 | 50 mg LY3053102 | 150 mg LY3053102 | 405 mg LY3053102 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 6
participants | 5 | 6 | 4 | 4 | 6 | 5 | 6

2. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Time Curve (AUC) of LY3053102
Description: AUC curve from time 0 to 168 hours postdose of LY3053102.
Time Frame: Time 0 to 168 hours after study drug administration on Day 1
Population: Participants who received at least one dose of LY3053102 and with evaluable LY3053102 concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour/milliliter
Groups:
- 2 mg LY3053102: LY3053102: A single dose of 2 mg, administered subcutaneously.
Arm/Group | 2 mg LY3053102 | 7 mg LY3053102 | 20 mg LY3053102 | 50 mg LY3053102 | 150 mg LY3053102 | 405 mg LY3053102
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6
microgram*hour/milliliter | 7.24 (29.6) | 16.1 (50.3) | 94.0 (45.5) | 192 (38.0) | 481 (74.0) | 1810 (49.1)

3. Secondary Outcome: PK: Observed Maximum Drug Concentration (Cmax) of LY3053102
Description: Cmax of LY3053102 from time 0 to 168 hours after study drug administration on Day 1.
Time Frame: Time 0 to 168 hours after study drug administration on Day 1
Population: Participants who received at least one dose of LY3053102 and with evaluable LY3053102 concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter
Arm/Group | 2 mg LY3053102 | 7 mg LY3053102 | 20 mg LY3053102 | 50 mg LY3053102 | 150 mg LY3053102 | 405 mg LY3053102
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6
microgram/milliliter | 0.0693 (30.2) | 0.140 (52.0) | 0.784 (46.8) | 1.68 (44.7) | 4.49 (67.6) | 16.2 (49.0)

4. Secondary Outcome: Number of Participants Who Developed Anti-LY3053102 Antibodies
Description: LY3053102 anti-drug antibodies (ADA) were assessed at baseline, 15 and 29 days. The number of participants with an initial postbaseline positive titer (defined as a >=2-fold increase in the ADA titer from baseline) anti-drug (LY3053102) ADA at each time point were summarized.
Time Frame: Baseline, up to Day 31
Population: Participants who received at least one dose of LY3053102 or placebo and with evaluable anti-drug (LY3053102) ADA data.
Measure: Number; unit: participants
Arm/Group | 2 mg LY3053102 | 7 mg LY3053102 | 20 mg LY3053102 | 50 mg LY3053102 | 150 mg LY3053102 | 405 mg LY3053102 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 6
participants
  Day 15 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Day 29 | 0 | 1 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | 2 mg LY3053102 | 7 mg LY3053102 | 20 mg LY3053102 | 50 mg LY3053102 | 150 mg LY3053102 | 405 mg LY3053102 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/5 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 5/6 | 6/6 | 4/6 | 4/5 | 6/6 | 5/6 | 6/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 mg LY3053102 (N=6) | 7 mg LY3053102 (N=6) | 20 mg LY3053102 (N=6) | 50 mg LY3053102 (N=5) | 150 mg LY3053102 (N=6) | 405 mg LY3053102 (N=6) | Placebo (N=6)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Injection site haematoma (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Temperature intolerance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural site reaction (Injury, poisoning and procedural complications) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 1 (3) | 2 (3) | 5 (6)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 2 (2) | 5 (5) | 4 (4) | 2 (2) | 5 (5) | 5 (5) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tobacco abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days